CLINICAL TRIAL: NCT00335621
Title: Replacement of Nebulised Ipratropium With Inhaled Tiotropium in Stable COPD
Brief Title: Replacement of Nebulised Ipratropium With Inhaled Tiotropium in Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated prior to recruitment - recruitment proved impossible
Sponsor: NHS Greater Glasgow and Clyde (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RN05RM001; REC 05/S0709/45; SSA 05/S0704/40
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2006-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; ipratropium; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: Inhaled Tiotropium

SUMMARY:
Some patients with chronic obstructive pulmonary disease (COPD) take nebulised treatments to ease the symptom of breathlessness, including the drug ipratropium. Nebulised bronchodilator drugs are taken up to 4 times through the day, and this can take up to 15 minutes each time. Although the treatment isbe effective, patients report that the time taken to set-up and use the nebuliser can be a disincentive to regular use. By contrast, an inhaler device is easy to use following appropriate instruction, and takes only a few seconds to administer. Inhaled tiotropium is a once daily treatment taken by inhaler which has been shown to be effective in COPD. We wish to assess whether inhaled Tiotropium as effective as nebulised ipratropium in patients with stable chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Tiotropium and ipratropium bromide are both antimuscarinic bronchodilators, licensed for the treatment of COPD with a similar side-effect profile. Tiotropium administered by an inhaler device (Handihaler®) has been shown to be superior to placebo and inhaled ipratropium bromide in patients with COPD, in both short term and longer term studies. The superiority of inhaled tiotropium over inhaled ipratropium bromide has been demonstrated for lung function tests and also for measures of health status. It is not known however if inhaled tiotropium is superior to ipratropium bromide administered via a nebuliser.

We wish to examine whether inhaled tiotropium is as effective and safe as nebulised ipratropium bromide in patients with chronic stable COPD.

Design The study will be a randomised, crossover study. The patients will not be blinded to the therapy but the technician performing the pulmonary function tests will be blinded to the patients' therapy.

Duration The length of the study for each patient will be 12 weeks.

Patient group Patients would be recruited from the population of patients supplied with a nebuliser from the respiratory department at Glasgow Royal Infirmary. Patients will be identified from those regularly attending the out-patients department and who have stable disease. Patients who frequently admitted to the respiratory ward with exacerbations of their disease will be excluded. Patients will be recruited at the rate of 2 per week. The study will be a single site study.

Following consent the patients would be asked to complete the St George's respiratory questionnaire, undergo brief spirometry and a general heath/satisfaction questionnaire, including the baseline and transitional dyspnoea index. Patient demographics will be collected including; age, sex, duration of COPD, smoking history, height, weight, concurrent therapy inhaled and oral.

The patients would then be randomised to either remain on their nebulised ipratropium for a further 6 weeks or to be commenced on inhaled tiotropium via the HandiHaler. Patients commenced on tiotropium would be given instruction on how to use the new inhaler and be told not to use their nebulised ipratropium. All other medication would remain the same. The patients randomised to ipratropium would be instructed on continue to take their nebulised ipratropium as before. All patients would be issued with a diary card on which they would record their pattern of nebuliser use, symptoms, adverse events and any additional medication required eg antibiotics. Patients will also be asked to record any health resource use, eg visits to their GP or admission to hospital on the diary card. A compliance check in the form of a capsule count will be undertaken.

At the end of the six weeks the patients would again undergo brief spirometry, and complete the St George's respiratory questionnaire and a general health/satisfaction questionnaire. At this point the patient's therapy will be crossed over, such that those who were taking the inhaler would now take the nebuliser and vice versa. There will be no wash out period between arms of the study, since comparisons will be made between baseline and the end of each period of treatment for lung function and questionnaires, and diary cards will be analysed only for the final 4 weeks of each treatment period. Those patients to commence on tiotropium would be given instruction on how to use their inhaler and those restarting ipratropium would be asked to take their nebulised therapy as before. All patients would be issued with a diary card on which they would record their pattern of nebuliser use, symptoms, adverse events and any additional medication required eg antibiotics. Patients will also be asked to record any health resource use, eg visits to their GP or admission to hospital on the diary card.

At the end of the second 6-week period the patients would again complete the St George's respiratory questionnaire, undergo brief spirometry and a general heath/satisfaction questionnaire as before. A compliance check in the form of a capsule count will be undertaken.

At the end of the study patients will be asked which therapy was preferred and a recommendation will be made to their GP depending on their preference.

Details of the patient's last dose of inhaled therapy will be recorded at the time of spirometry.

Patient numbers The number of patients to be included in the study is 45. The patient numbers are based on a 90% statistical power to detect a mean change of 0.2L in FEV1 between visits 2 and 3 as a result of treatment, using a 5% significance level paired test. This justification is based on previous studies which conservatively indicate the standard deviation of FEV1 values to be 0.4L. Statistical analysis will be undertaken for differences in the mean FEV1 values between visits 2 and 3 using a paired design and parametric testing. Results will be presented using the differences in means between treatments and the associated 95% confidence interval. Other response variables will be similarly analysed for evidence of any difference in treatment effect, with analysis of diary cards only for the final 4 weeks of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stable Moderate to severe COPD (GOLD criteria)
* > 20 pack year smoking history
* current treatment with nebulised ipratropium bromide
* no exacerbations within preceding 3 months

Exclusion Criteria:

* current participation in other study
* < 20 pack year smoking history
* Significant co-morbidity e.g. cardiac
* history of intolerance to lactose

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-06; Study Completion 2007-12

PRIMARY OUTCOMES:
Spirometry

SECONDARY OUTCOMES:
St George's Respiratory Questionnaire
Baseline/Transition Dyspnea index

CONTACTS AND LOCATIONS:
Overall Officials: George W Chalmers, MD, Principal Investigator — NHS Greater Glasgow and Clyde; Anne Boyter, PhD, Principal Investigator — Strathclyde University
Locations (1):
- Department of Respiratory Medicine, Glasgow Royal Infirmary, Glasgow, United Kingdom